CLINICAL TRIAL: NCT04669951
Title: Urokinase-type Plasminogen Activator Receptor and Gastroesophageal Adenocarcinomas
Brief Title: Urokinase-type Plasminogen Activator Receptor and Gastroesophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Patrick Achiam (Other)
Responsible Party: Sponsor-Investigator, Michael Patrick Achiam, Consultant, MD, DMSci, Ph.D., FEBS-OG, Ass. Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: uPAR ECV
Record Dates: First submitted 2020-12-02; First posted 2020-12-17 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Esophagus Cancer, Adenocarcinoma
Keywords: urokinase plasminogen activator receptor; uPAR; Cardia; Adenocarcinoma; Immunohistochemistry
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: The patients will be drawn from the existing clinical biobank. The biobank is located at the department of pathology, Rigshospitalet. From this clinical biobank, a new temporary research biobank will be made. Supplementary sections from formalin-fixed paraffin embedded (FFPE) blocks containing tumor tissue will be cut and Haematoxylin and eosin (HE) and immunohistochemical (IHC) staining will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- uPAR expression (Experimental): Immunohistochemistry
  Interventions: Other: uPAR immunohistochemistry

INTERVENTIONS:
Other: uPAR immunohistochemistry — Resected esophageal cancer will be qualitatively and semi-quantitatively analyzed for uPAR expression

SUMMARY:
The aim of this study is to investigate urokinase Plasminogen Activator Receptor (uPAR) microexpression in gastroesophageal cancer (adenocarcinomas) both qualitatively and semi-quantitatively and to evaluate if it offers a possibility for future imagining purposes.

DETAILED DESCRIPTION:
* Sections of the tumor tissue will be HE stained.
* Sections of the tumor tissue will be stained with an uPAR antibody for immunohistochemistry.
* Immunohistochemical staining against cytokeratin which colors cancer cells will be made to assist the observer in the evaluation of uPAR microexpression pattern.
* A semiqualitative scale corresponding to the level of uPAR expression will be made.
* Quantitative polymerase chain reaction will be used to validate the immunohistochemistry uPAR expression pattern.
* An electronic scoring system (digital pathology) will be trained to access the expression of uPAR in both tumor- and normal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Patients who underwent curatively intended surgery for gastroesophageal cancer
* Patients who underwent surgery after 01-01-2016.

Exclusion Criteria:

* Patients who applied for an exception from medical research at the "National Registry of Tissue Use."
* Patients with other histological subtypes than adenocarcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
uPAR microexpression | Up to 6 months
  Our primary objective is to investigate uPAR microexpression in gastroesophageal adenocarcinomas both qualitatively and semi-quantitatively. This will be done by a pathology analysis of gastroesophageal cancer resections.
Tumor-to-background ratio | Up to 6 months
  A pathology staining will determine the uPAR in the tumor compared with the healthy cells.

SECONDARY OUTCOMES:
uPAR in patient groups | Up to 6 months
  Baseline statistical analysis of patient groups and their expression of uPAR in their resected tumor tissues will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Achiam, MD., Ph.D, Principal Investigator — Rigshospitalet, Department of Surgical Gastroenterology
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark